CLINICAL TRIAL: NCT03671421
Title: Number One Overall Graft Pick? Hamstring vs Bone-Patellar-Tendon-Bone vs Quadriceps Tendon: A Prospective Cohort Study
Brief Title: Number One Overall Graft Pick? Hamstring vs Bone-Patellar-Tendon-Bone vs Quadriceps Tendon
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Department head, orthopaedic surgery, Panam Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2016:066
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Graft choice; hamstring; quadriceps tendon
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Prospective quasi-randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The clinical assessments will be done by someone blinded to the arm of the study the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quads tendon (Active Comparator): The graft tissue will be quadriceps tendon
  Interventions: Procedure: ACL reconstruction - graft choice
- Hamstring (Active Comparator): Semitendinosus and gracilis will be used for graft
  Interventions: Procedure: ACL reconstruction - graft choice
- BPTB (Active Comparator): Bone patellar tendon bone graft to be used.
  Interventions: Procedure: ACL reconstruction - graft choice

INTERVENTIONS:
Procedure: ACL reconstruction - graft choice — Use of 3 different ipsilateral autograft options

SUMMARY:
The main purpose of this study is to determine if there is a difference in graft re-injury/failure rates between participants that have had an ACL reconstruction with a STG, BPTB or QT autograft. Additionally, to compare quality of life, patient reported outcomes and functional performance after ACL reconstruction with STG, BPTB and QT.

DETAILED DESCRIPTION:
The main purpose of this study is to determine if there is a difference in graft re-injury/failure rates between participants that have had an ACL reconstruction with a STG, BPTB or QT autograft. Additionally, to compare quality of life, patient reported outcomes and functional performance after ACL reconstruction with STG, BPTB and QT.

Quasi-randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* - confirmed diagnosis of a complete primary unilateral ACL rupture based on all of the following:
* history of a traumatic injury episode
* physical exam findings of increased anterior translation of the tibia on the femur (Lachman test and/or anterior drawer test)
* positive pivot shift test
* patients must be 14 to </= 50 years (at time of surgery)
* x-rays showing skeletal maturity (i.e. tibial tubercle fused) and no fractures
* MRI prior to surgery (note: if the radiologist's report states an incomplete or partial ACL on MRI but the surgeon diagnoses the patient with a complete unilateral tear based on the clinical criteria above, then the patient will be considered eligible. Final eligibility will be determined intra-operatively.)

Exclusion Criteria:

* - ACL rupture on contra-lateral limb
* Partially torn ACL *final determination made intra-operatively
* Concomitant medial collateral, lateral collateral, or posterior collateral ligament tears requiring surgical repair *final determination made intra-operatively
* Severe chondromalacia (Grade IV on the ICRS scale) *final determination made intra-operatively
* ACL reconstruction using allograft tissue
* Confirmed connective tissue disorder
* Unwillingness to be followed for 24 months post-operatively
* History of rheumatoid arthritis
* Pregnancy (at the time of surgery)
* Psychiatric illness that precludes informed consent
* Unable to speak, read or understand the English language
* Major medical illness (life expectancy less than 1 year or unacceptably high operative risk)

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 297 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
graft re-injury (re-rupture, partial tear) or graft failure | 24 months
  ) Diagnosis of a complete graft re-rupture requires all of the following criteria to be met:
  * associated with an acute traumatic event
  * a definite loss of end point on manual Lachman testing
  * increased anterior translation >3 mm
  * > or = Grade 2 pivot shift
  * tear confirmed as complete on MRI or diagnostic arthroscopy
  * revision ACL reconstruction IS recommended or required
    2) Diagnosis of a partial re-rupture requires all of the following criteria:
  * suspected meniscal injury or graft tear on history without the clinical characteristics of a complete rupture
  * tear confirmed as partial by MRI or diagnostic arthroscopy
  * revision ACL reconstruction is NOT recommended or required
    3) Diagnosis of graft failure will be defined as:
  * >/= Gr. 2 pivot shift and/or >6 mm side-to-side difference on manual Lachman

SECONDARY OUTCOMES:
SANE | 24 months
Knee laxity | 24 months
  KT1000 Knee Laxity Arthrometer
Concentric maximal strength | 24 months
  Knee flexion and extension strength - biodex
Pain log | 3 weeks post operative
  type and quantity of pain medication use
ACL-QOL | 24 months
SF-12 | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No